CLINICAL TRIAL: NCT02673879
Title: A Trial of Complete Percutaneous Pericardial Drainage Facilitated by Intrapericardial Alteplase Compared to Conventional Pericardiocentesis When Indicated in Adults With Large Pericardial Effusion Due to Tuberculous and Non-tuberculous Pericarditis
Brief Title: IMPI 2 - A Trial of Intrapericardial Alteplase in Large Pericardial Effusion
Acronym: IMPI-2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cape Town (Other)
Collaborators: Walter Sisulu University (Other); Population Health Research Institute (Other)
Responsible Party: Principal Investigator, Bongani M Mayosi, Professor of Medicine, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HREC REF No. 370/2015
Record Dates: First submitted 2016-02-01; First posted 2016-02-04 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2016-02

CONDITIONS: Pericardial Effusion
MeSH Terms: conditions — Pericardial Effusion | interventions — Pericardiocentesis; Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pericardiocentesis with Alteplase (Active Comparator): Complete percutaneous pericardial drainage facilitated by intrapericardial alteplase.
  Interventions: Other: Pericardiocentesis with Alteplase
- Conventional Pericardiocentesis (Other): Conventional pericardiocentesis when indicated.
  Interventions: Other: Conventional Pericardiocentesis

INTERVENTIONS:
Other: Pericardiocentesis with Alteplase — Complete percutaneous pericardial drainage facilitated by intrapericardial alteplase
  Arms: Pericardiocentesis with Alteplase
Other: Conventional Pericardiocentesis — Conventional pericardiocentesis when indicated
  Arms: Conventional Pericardiocentesis

SUMMARY:
The Second Investigation of the Management of Pericarditis (IMPI-2) Trial will compare the effectiveness and safety of complete percutaneous pericardial drainage facilitated by intrapericardial alteplase (recombinant human tissue-type plasminogen activator) to conventional pericardiocentesis when indicated in 2176 patients with large pericardial effusion due to tuberculous and non-tuberculous pericarditis. An internal pilot study of 218 patients will initially confirm the feasibility of conducting a large-scale multi-centre clinical trial of intrapericardial fibrinolysis in patients with large pericardial effusion, and also provide preliminary safety data, following a dose finding study of intrapericardial alteplase.

DETAILED DESCRIPTION:
Intrapericardial fibrinolytic agents are used in the drainage of tuberculous, purulent, neoplastic and other inflammatory pericardial effusions to prevent recurrent effusions and constrictive pericarditis. This use is based on evidence from case reports and a small trial that did not have the statistical power to reliably evaluate the effect of pericardial drainage facilitated by intrapericardial fibrinolysis on safety and important clinical outcomes.

The Second Investigation of the Management of Pericarditis (IMPI-2) Trial will compare the effectiveness and safety of complete percutaneous pericardial drainage facilitated by intrapericardial alteplase (recombinant human tissue-type plasminogen activator) to conventional pericardiocentesis when indicated in 2176 patients with large pericardial effusion due to tuberculous and non-tuberculous pericarditis. An internal pilot study of 218 patients will initially confirm the feasibility of conducting a large-scale multi-centre clinical trial of intrapericardial fibrinolysis in patients with large pericardial effusion, and also provide preliminary safety data, following a dose finding study of intrapericardial alteplase.

Hypothesis: We hypothesise that patients with large pericardial effusion randomized to intrapericardial alteplase to ensure complete pericardial drainage will have at least a 35% reduction in cardiac tamponade requiring pericardiocentesis or constrictive pericarditis compared to conventional pericardiocentesis when indicated.

Objectives: The primary objectives of the IMPI-2 Trial are:

1. To demonstrate the feasibility of conducting a multicentre clinical trial of intrapericardial fibrinolysis in patients with large pericardial effusion, and to assess the safety of intrapericardial alteplase in an internal pilot study, and
2. To determine the effectiveness of intrapericardial alteplase in reducing the composite outcome of cardiac tamponade requiring pericardiocentesis or constrictive pericarditis in patients with large pericardial effusion in the full trial.

Should the internal pilot study demonstrate feasibility and safety; all 218 patients will be rolled-over into the full scale IMPI-2 trial of 2176 participants. The primary outcome is the first occurrence of cardiac tamponade requiring pericardiocentesis or constrictive pericarditis. The secondary safety endpoint is safety of intrapericardial fibrinolysis measured by effect on major bleeding, and serious and non-serious adverse events. The secondary efficacy outcomes are constrictive pericarditis, and cardiac tamponade requiring pericardiocentesis, analysed separately, and persistent or recurrent pericardial effusion without cardiac tamponade, hospitalisation, and death. The secondary diagnostic outcomes are proportion with bacteriologically confirmed tuberculosis from any organ or tissue; time to diagnosis of bacteriologically confirmed tuberculosis in days; accuracy of novel tests for the diagnosis of tuberculosis; proportion with specific diagnosis of any pericardial disease; time to diagnosis of a specific pericardial disease in days.

Study Design: IMPI-2 is a prospective randomized open blinded end-point trial that will enroll 2176 patients with large pericardial effusion over 36 months from up to 30 centres in South Africa and Africa. Eligible patients will be randomly assigned to receive complete pericardial drainage facilitated by intrapericardial fibrinolysis or conventional pericardiocentesis when indicated on enrollment to the study. Patients will be followed at 2 weeks, 6 weeks, 12 weeks, and in months 6, and 12 after enrollment. The IMPI Project Office, University of Cape Town, South Africa will manage and coordinate the study in association with the Pericarditis Research Unit, Walter Sisulu University, South Africa and the Population Health Research Institute, McMaster University, Canada.

Importance: IMPI-2 addresses very serious complications of large pericardial effusion (i.e., cardiac tamponade and constrictive pericarditis), which are associated with high mortality despite pericardiocentesis or pericardiectomy. This study will utilise the research network that was established by the IMPI trial which was completed in 2014.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age;
2. Confirmed large pericardial effusion on echocardiography (i.e., echo free space ≥1 cm anterior to the right ventricle of the heart in diastole);
3. Willingness to participate for the full duration of the trial (i.e., 12 months); and
4. Provision of written informed consent.

Exclusion Criteria:

1. Age < 18 years;
2. Uraemic pericarditis (i.e., urea > 21.4 mmol/l);
3. Thrombocytopenia (i.e., < 100,000 platelets per µl);
4. Presence of a contra-indication to the administration of a fibrinolytic agent (i.e., major haemorrhage or major trauma; coincidental stroke; major surgery in the previous 5 days; blood pressure >200/100 mmHg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2176 (Estimated)
Dates: Start 2016-02; Primary Completion 2019-07 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Composite outcome of cardiac tamponade requiring pericardiocentesis or constrictive pericarditis. | 12 months
  Cardiac tamponade requiring pericardiocentesis shall refer to a combination of physical and echocardiographic findings, i.e., patients with clinical signs of tachycardia (> 90 bpm), hypotension (systolic blood pressure < 100 mmHg), elevated jugular venous pressure and/or pulsus paradoxus > 10 mmHg plus evidence of a large pericardial effusion with echocardiographic signs of tamponade in the absence of other cardiac disease, as defined in the IMPI trial.
  Constrictive pericarditis shall refer to a combination of physical and echocardiographic findings (i.e., patients with a prior history of pericardial effusion who have pulsus paradoxus, a raised jugular venous pressure with or without evidence of pericardial thickening on imaging) in the absence of either large pericardial effusion or other cardiac disease, as described in the IMPI trial.

SECONDARY OUTCOMES:
Major bleeding | 12 months
  Defined as clinically overt bleeding accompanied by one or more of the following: a decrease in the haemoglobin level of 2 g per decilitre or more over a 24-hour period, transfusion of 2 or more units of packed red cells, bleeding at a critical site (intracranial, intraspinal, intraocular, pericardial, intraarticular, intramuscular with compartment syndrome, or retroperitoneal), or fatal bleeding
Clinically relevant non-major bleeding | 12 months
  Defined as clinically overt bleeding that does not satisfy the criteria for major bleeding and that leads to hospital admission, physician-guided medical or surgical treatment.
Any bleeding | 12 months
  Any other form of bleeding that is not covered by safety outcomes 1-3
Other adverse events | 12 months
  Any other adverse events
Persistent pericardial effusion without cardiac tamponade | 12 months
  Refers to the echocardiographic presence of a pericardial effusion without criteria for cardiac tamponade requiring pericarditis during follow-up visits. The pericardial effusion is the same size or larger than that measured at the time of enrollment (where no pericardiocentesis was done) or post-pericardiocentesis.
Recurrent pericardial effusion without cardiac tamponade | 12 months
  Refers to the echocardiographic presence of a pericardial effusion without criteria for cardiac tamponade requiring pericarditis during follow-up visits. Recurrence is present in the context of re-appearance of a pericardial effusion in the context where complete drainage was performed.
Hospitalisation for any cause; and death from any cause | 12 months
  Refers to admission to hospital for at least 24 hours for any reason.
Cardiac tamponade requiring pericardiocentesis | 12 months
  Cardiac tamponade requiring pericardiocentesis shall refer to a combination of physical and echocardiographic findings, i.e., patients with clinical signs of tachycardia (> 90 bpm), hypotension (systolic blood pressure < 100 mmHg), elevated jugular venous pressure and/or pulsus paradoxus > 10 mmHg plus evidence of a large pericardial effusion with echocardiographic signs of tamponade in the absence of other cardiac disease, as defined in the IMPI trial.
Constrictive pericarditis | 12 months
  Constrictive pericarditis shall refer to a combination of physical and echocardiographic findings (i.e., patients with a prior history of pericardial effusion who have pulsus paradoxus, a raised jugular venous pressure with or without evidence of pericardial thickening on imaging) in the absence of either large pericardial effusion or other cardiac disease, as described in the IMPI trial.
Death | 12 months
  Death from any cause

OTHER OUTCOMES:
Proportion with proven tuberculosis | 12 months
  The proportion with bacteriologically confirmed tuberculosis from any organ or tissue in each group will be based on findings on microscopy, Xpert MRB/RIF, culture, and / histology .
Time to diagnosis of proven tuberculosis | 12 months
  The time to diagnosis of bacteriologically confirmed tuberculosis in days in each group will be based on the date of sample collection and the date of first bacteriological confirmation from any organ or tissue.
Proportion with proven tuberculosis on novel tests who are not put on treatment | 12 months
  The proportion of culture-positive tuberculosis cases who are not placed on treatment in either arm, or the proportion of these which would have been detected by the novel rapid index tests.
Diagnostic accuracy of novel tests of tuberculosis | 12 months
  The diagnostic accuracy of novel tests (e.g., Xpert MTB/RIF, Xpert ULTRA, InterGam) for the detection of culture-positive pericardial tuberculosis (a secondary analysis will be performed using clinically-diagnosed tuberculosis as reference standard)
Drug resistant tuberculosis | 12 months
  The proportion of drug-resistant tuberculosis cases detected.
Specific diagnosis of tuberculous pericarditis | 12 months
  The proportion with a specific diagnosis of pericardial disease in each group will be based on findings on results of investigations for tuberculosis, cancer, purulent pericarditis and other disease.
Time to diagnosis of specific pericardial disease | 12 months
  The time to diagnosis of a specific pericardial disease in days in each group will be based on the date of sample collection and the date of first definitive result.

CONTACTS AND LOCATIONS:
Overall Officials: Bongani M Mayosi, DPhil, Principal Investigator — University of Cape Town
Locations (1):
- Groote Schuur Hospital, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data will be made available on request at the end of the study, subject to approval by the Steering Committee of the IMPI-2 Trial.